CLINICAL TRIAL: NCT05775627
Title: Uncovering Sleep and Circadian Mechanisms Contributing to Adverse Metabolic Health
Brief Title: Sleep and Metabolism
Acronym: SAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00025152
Record Dates: First submitted 2022-11-18; First posted 2023-03-20 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Sleep Deprivation; Obesity; Glucose Intolerance; Weight Gain; Food Selection
Keywords: sleep restriction; obesity; glucose intolerance; weight gain; circadian timing; ad libitum; food selection
MeSH Terms: conditions — Sleep Deprivation; Obesity; Glucose Intolerance; Weight Gain; Food Preferences

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction First (Experimental): Equivalent to obtaining 5.5.h of sleep per 24h; n=10. Participants live on a 20h-day and will experience 15.33h wake episodes followed by sleep episodes of 4.67h long.
  Ad libitum food is provided during this time and participants will be fed ~130-150% of their daily caloric needs across three meals a day.
  Interventions: Behavioral: Sleep Restriction
- Controlled Condition First (No Intervention): Equivalent to obtaining 8h sleep per 24h; n=10. Participants live on a 20h-day and will experience 13.33h wake episodes followed by 6.67h sleep opportunities.
  Ad libitum food is provided during this time and participants will be fed ~130-150% of their daily caloric needs across three meals a day.

INTERVENTIONS:
Behavioral: Sleep Restriction — Participants are randomized into either a group (n=10) that is sleep restricted first or control first (n=10) group; the groups will crossover halfway through the protocol. Both arms are fed 3 meals and have access to ad libitum food between meals. Both groups will also undergo up to 3 mixed-meal tolerance tests to measure glucose tolerance.
  Arms: Sleep Restriction First

SUMMARY:
The goal of this study is to uncover sleep and circadian mechanisms contributing to adverse metabolic health. The protocol is a 21 day (7 outpatient days, 14 inpatient days) mechanistic randomized-crossover study designed to identify the impact of chronic sleep restriction and circadian timing, independently and in combination on energy metabolism and identify the independent and combined effects on glucose tolerance.

DETAILED DESCRIPTION:
Nearly half of all Americans are obese and/or have been diagnosed with diabetes, accounting for over 327 billion dollars in health care costs in the United States each year. Increasing evidence suggests that chronic short-sleep durations contribute to these diseases, but the specific mechanisms as to how short-sleep durations results in weight gain and diabetes are debated.

Reports of weight gain due to sleep restriction do not comply with the energy balance hypothesis, which would predict that with an increased amount of wakefulness and an associated increase in energy expenditure, there would be a negative shift in energy balance and resulting weight loss over time. Restricting sleep in the laboratory, however, pushes participants towards a positive energy balance via increased daily energy intake when access to food is ad libitum.

The goals of this study are to uncover the impact of chronic sleep restriction, circadian timing, and their combination on energy intake patterns, determine the influence of chronic sleep restriction on food choice when there is equal opportunity to eat at all circadian times, and discover the impact of chronic sleep restriction, circadian timing, and their combination, on glucose tolerance.

1. Ambulatory monitoring: Participants will maintain a consistent 7-day at home 8h sleep schedule at habitual times before both laboratory visits to ensure 1) subjects are not sleep restricted and 2) that they are obtaining the same light-dark schedule prior to each laboratory visit for stable entrainment; verified by actigraphy, sleep logs, and call-ins to a time stamped recorder. Drugs, medications, caffeine, alcohol, and nicotine will be prohibited to use during this time and toxicology analysis will be performed upon admission.
2. Outpatient diet: For 3-days prior to each protocol, participants will consume an outpatient isocaloric diet designed to meet individual daily energy requirements. The diet will consists of a breakfast, lunch, dinner, and snack and participants will be trained by staff in how to prepare the meals. Participants will be instructed to only consume the food provided during these 3-days and be asked by staff to confirm this is all they ate via daily check-ins to ensure adherence.
3. Inpatient protocols: Participants will be admitted to an individual room free of external time cues (e.g. clocks, radios, computers, visits and sunlight). Room temperature is maintained at 21 - 22.2 degrees Celsius and light intensity set at ≤5 lux during forced desynchrony procedures and 0 lux (darkness) during scheduled sleep opportunities. Participants will be instrumented for full polysomnography (PSG) and given a telemetry pill for continuous core body temperature measurement. An 18-gauge IV catheter will also be inserted into the forearm and connected to a triple-stopcock manifold via an IV loop with a 12-foot small-lumen extension cable through which blood sampling can continue in the next room without disturbing leisure activity or sleep.

After instrumentation, participants will be given an 8h sleep opportunity at habitual timing (determined via actigraphy) and will be awakened at habitual wake time in dim-lighting for a baseline "day". During baseline, participants will be given three energy-balanced meals. After baseline, participants' sleep/wake schedule will be advanced by 4h daily for the next 12 calendar days with the participants having access to ad libitum food. Prior to arriving to the laboratory, participants will be randomized to either sleep restriction first (equivalent to obtaining 5.5h of sleep per 24h; n=10) or control conditions first (equivalent to 8h sleep per 24h; n=10); crossover to the other condition will occur on day 8 of the protocol. Because the protocol requires participants to live on a 20h-day, during the control condition participants will experience 13.33-hour wake episodes followed by 6.67-hour sleep opportunities, while during the sleep restriction condition they will experience 15.33-hour wake episodes followed by sleep episodes of 4.67 hours long, in the range typically experienced by individuals who habitually restrict their sleep. Providing ad libitum food during this time will be accomplished, as done previously, by providing participants a breakfast, lunch and dinner at ~130-150% more calories than their baseline day and switching out sets of snacks between meals - "morning" (between breakfast and lunch), "afternoon" (between lunch and dinner), and after-dinner (between dinner and sleep). Snacks will be of a variety of healthy (i.e., grapes, low-fat yogurts, whole-grain crackers, nuts, etc.) and unhealthy (i.e., ice cream, cookies, chips, sodas, etc.) options and participants will not need to ask or record what they eat.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age
* Drug free
* Established disease-free status

Exclusion Criteria:

1. Dietary restrictions

   Participants must not have dietary restrictions that could systematically bias their macronutrient intake. The following will exclude participants from enrolling in the study based on their diet:
   * Participants who choose not to or cannot consume dairy products (milk, yogurt, cheese, ice cream)
2. Body Composition

   A body mass index (BMI) of 18.5< [BMI] < 25 kg/m2 and a waist circumference <94/80cm.
3. Psychiatric/psychological suitability

   Each participant will undergo a structured interview (Mini International Neuropsychiatric Interview) with a qualified OHSU physician. This physician will supervise the administration and scoring of a Beck Depression Inventory II (BDI-II) questionnaire for each potential participant. The following will exclude individuals from participating based on their psychiatric or psychological evaluation:
   * Individuals with evidence of psychopathology on the BDI-II, or in a structured clinical interview with the physician
   * A history of severe psychiatric illnesses
   * Alcoholism
   * Drug dependency
   * Major depression
   * Manic depressive illness
   * Schizophrenic disorders
   * Panic disorder
   * Generalized anxiety disorder
   * Post-traumatic stress disorder
   * Agoraphobia
   * Claustrophobia
   * Paranoid personality disorder
   * Schizoid personality disorder
   * Schizotypal personality disorder
   * Borderline personality disorder
   * Antisocial personality disorder.
   * History of using antidepressant medication
   * History of using neuroleptic medication
   * History of using tranquilizers
4. Drug/alcohol use

   Volunteers must be drug-free (including caffeine, nicotine, alcohol and herbal medications) for the entire duration of the outpatient and in-laboratory study period, with no history of drug or alcohol dependency. All participants must be:
   * Current non-smokers, and are required to have a history of less than 5 'pack years' of smoking
5. Medication/drug use

   Volunteers must not be taking any prescribed medications or over the counter medications, with an exception for birth control.
6. Prior shift work

   For stability of endogenous circadian rhythmicity, volunteers must have no history of the following 1 year prior to the study:
   * Working irregular day and night hours
   * Regular night work
   * Rotating shift work f
   * Not have traveled more than 1 time zone during 3 months prior to the study
7. Chronobiologic and sleep disorders

   * Hypernychthemeral sleep/wake cycle
   * Delayed sleep phase syndrome (wake time > 2 hours later than desired or habitually after 10:00 AM)
   * Advanced sleep phase syndrome (wake time > 2 h earlier than desired or habitually before 5:00 AM)
   * Narcolepsy
   * Sleep apnea (apnea index >15)
   * Insomnia (sleep complaint by history or polygraphically recorded sleep efficiency < 80%)
   * Hypersomnia
   * Periodic Limb Movement (PLMS) (PLMS index >15)
   * Nocturnal Paroxysmal Dystonia
   * REM-sleep behavior disorder
   * Nocturnal Enuresis; (self-report and first night in the laboratory)
   * Obstructive sleep apnea (apnea/hypopnea index >5/h as determined by at-home monitoring)
   * The investigators will also exclude individuals with extreme chronotype using the Horne-Ostberg Morningness/Eveningness questionnaire (i.e., the Owl/Lark Questionnaire)
8. Diseases of the Cardiovascular System

   * Hypertension (systolic blood pressure > 140 or diastolic blood pressure > 90)
   * Heart failure
   * Cardiomyopathy
   * Cor pulmonale
   * Ischemic heart disease
   * Valvular heart disease
   * History of heart transplantation
   * Cardiac tumors
   * Pericardial disease
9. Metabolic Syndrome

   Following American Heart Association cutoffs, participants who have, in addition to abdominal fat (obese exclusion criteria), two or more of these factors will be excluded from the study:
   * HDL cholesterol of less than 40 mg/dL in men or less than 50 mg/dL in women
   * Systolic blood pressure >135 mmHg or diastolic blood pressure >85 mmHg
   * Fasting blood glucose ≥ 100 mg/dL
   * Triglycerides ≥ 150 mg/dL
10. Pre-Diabetes/Diabetes

    For participants who have a fasting blood glucose level of ≥ 100 mg/dL the investigators will measure hemoglobin A1c to exclude for diabetes (HbA1c>5.7%).
11. Hypertension

    An upper cut off of 140/90 mmHg during an office blood pressure measure will be used as an exclusion criterion. After 5 minutes of rest in a seated position, blood pressure will be measured 3 times, taken 1 minute apart. The average will be used to confirm eligibility criteria. Current or history of beta blocker use will also be exclusionary.
12. Disorders of the Respiratory System

    * Asthma
    * Cystic fibroses
    * Chronic bronchitis
    * Emphysema
    * Airway obstruction
    * Interstitial lung diseases
    * Pulmonary hypertension
    * Lung neoplasms
    * ARDS
13. Disorders of the Kidney and Urinary Tract

    * Acute or chronic renal failure
    * History of renal transplantation
    * Tubulointerstitial diseases of the kidney
    * Urinary tract obstruction
    * Tumors of the urinary tract
14. Infectious Diseases

    * Infective endocarditis
    * HIV infection
    * Sexually transmitted diseases [e.g., syphilis (including congenital syphilis and its sequelae), gonorrhea],
    * Urinary tract infection
    * Osteomyelitis
    * Brucellosis
    * Toxoplasmosis,
    * Tuberculosis
    * Leptospirosis
    * Lyme disease
    * Mononucleosis
    * Hepatitis
    * Parasitic infections such as malaria, toxoplasmosis, giardiasis, schistosomiasis, leishmaniasis
15. Disorders of the Gastrointestinal System

    * Esophagitis
    * Peptic ulcer and gastritis
    * Neoplasms of the esophagus, stomach or bowel
    * Disorders of absorption
    * Inflammatory bowel disease
    * Diseases of the small and large intestine
    * Acute appendicitis
    * Cirrhosis or neoplasms of the liver
    * History of liver transplantation
    * Diseases of the gallbladder and bile ducts
    * Pancreatic disease
16. Disorders of the Immune System, Connective Tissue and Joints

    * AIDS
    * Systemic lupus erythematosus
    * Rheumatoid arthritis
    * Scleroderma
    * Ankylosing spondylitis
    * Vasculitis
    * Sarcoidosis
17. Disorders of the Hematopoietic System

    * Anemia
    * Leukemia
    * Myeloproliferative diseases
    * History of bone marrow transplantation
18. Neoplastic Diseases

    * Lymphoma
    * Carcinoma
    * Melanoma
    * Any other neoplastic diseases
19. Endocrine and Metabolic Diseases

    * Thyroid disease
    * Addison's Disease
    * Cushing's Syndrome
    * Aldosteronism
    * Hypoaldosteronism
    * Pheochromocytoma
    * Disorders of sexual differentiation that require hormone supplementation that may alter body weight
    * Disorders of neuroendocrine regulation
    * Diseases of the anterior pituitary and hypothalamus
    * Hemochromatosis porphyria
    * Wilson's Disease
    * Glycogen storage diseases
    * Diseases of the parathyroid gland
    * Metabolic bone disease
    * Disorders of phosphorus or magnesium metabolism
    * Paget's Disease
20. Neurologic Disorders

    * Epilepsy and disorders of consciousness
    * Dementia
    * Amnesic disorders
    * Neoplastic diseases of the central nervous system
    * Demyelinating diseases
    * Parkinson's Disease
    * Muscular dystrophy
    * Myasthenia gravis
    * Periodic paralysis
    * Dermatomyositis
    * Polymyositis
    * Infections of the nervous system
    * Stroke
    * History of transient ischemic attacks
    * Hydrocephalus
    * Tumors of the pituitary gland
    * Pinealoma
    * Intervertebral disc disease
    * Ataxia
    * Gilles de la Tourette Syndrome
    * Huntington's Disease
    * Tardive dyskinesia
    * History of recurrent migraine headaches
    * Neuromuscular disease.
21. Subjects must not be currently participating in another research study that would influence their safe participation in our study. Subjects must not be participating in a research study in which they do the following:

    * Ingest experimental medication
    * Give blood samples

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Circadian Phase | 14 days
  Saliva will be assayed for melatonin used standardized assays. Melatonin will be sampled at 1h intervals during wakefulness. Melatonin onset will be calculated using the linear interpolated time at which melatonin levels reach 25% of a fitted peak-to-trough amplitude.
Energy Intake | 14 days
  Throughout the forced desynchrony protocol, participants will have ad libitum access to food, which will be scored using NDSR software. NDSR was developed to help plan, manage, and analyze food and nutrient intake. Each meal and set of snacks will be timestamped (midpoint of snack availability) and binned by circadian phase based on the individuals' melatonin and also by time awake.
Energy Content | 14 days
  Throughout the forced desynchrony protocol, participants will have ad libitum access to food, which will be scored using NDSR software. NDSR was developed to help plan, manage, and analyze food and nutrient intake. Each meal and set of snacks will be timestamped (midpoint of snack availability) and binned by circadian phase based on the individuals' melatonin and also by time awake.
Glucose Metabolism | ~3 days
  The participant's glucose and insulin response to a mixed meal diet high in carbohydrates may be tested up to 3 times during the protocol (Days 2, 4, and 13). Each participant will have a choice of 1 of 2 meal options and will be given that meal throughout the study. During this mixed meal test, a baseline blood draw will occur ~7-min before the meal and then the frequency of blood samples will increase to every 10-min after the meal for 90 min and then every 30 min for 90 min for a total of 14 samples (~1 mL each, total of ~14 mL) over 180 minutes to measure glucose and hormone response in detail. Samples at each time point will be obtained for measurement of suppressibility of plasma free fatty acids. Blood will also be drawn every 4h during the protocol for 24h insulin and glucose.
Resting energy expenditure | 14 days
  Resting energy expenditure will be measured upon awaking each protocol day via indirect calorimetry. Oxygen consumption and carbon dioxide production will be used to calculate metabolic rate.
Resting energy macronutrient oxidation | 14 days
  Resting macronutrient oxidation will be measured upon awaking each protocol day via indirect calorimetry. Oxygen consumption and carbon dioxide production will be used to calculate the oxidation of carbohydrate and fat.
Blood Pressure | 14 days
  Beat-to-beat blood pressure will be obtained using a non-invasive device employing the volume-clamp method with hydrostatic correction (Nexfin). Beat-to-beat blood pressure will be recorded 1) during each sleep episode and 2) each constant posture period following awakening. Both systolic and diastolic blood pressure will be measured.
Heart Rate | 14 days
  For the duration of the study, 2 channels of EKG are recorded (RA-V6) and stored on BioPac recorders using Acqknowledge software (256 Hz).
Sympathetic Activity | 14 days
  The investigators will use the high frequency power of the heart rate variability power spectrum to estimate cardiac parasympathetic activity (vagal tone) as modulated by respiratory sinus arrhythmia. RR interval data for sequential 5-minute time segments will be used for heart rate variability analysis according to published criteria. Frequency domain measures are calculated by interpolating the RR tachogram with a cubic spline and re-sampling. Power spectral density will be calculated using Welch's technique. Calculated time domain heart rate variability measures will include mean RR, SD of all normal-normal RR intervals, and a percentage of RR intervals differing by greater than 50 msec.
Parasympathetic Activity | 14 days
  The investigators will use the high frequency power of the heart rate variability power spectrum to estimate cardiac parasympathetic activity (vagal tone) as modulated by respiratory sinus arrhythmia. RR interval data for sequential 5-minute time segments will be used for heart rate variability analysis according to published criteria. Frequency domain measures are calculated by interpolating the RR tachogram with a cubic spline and re-sampling. Power spectral density will be calculated using Welch's technique. Calculated time domain heart rate variability measures will include mean RR, SD of all normal-normal RR intervals, and a percentage of RR intervals differing by greater than 50 msec.
Vascular Endothelial Function | 14 days
  The investigators will measure vascular endothelial function at various points throughout the protocol. Brachial or femoral artery flow-mediated dilation will be measured in the supine position.
Leptin | 14 days
  The investigators will measure markers of hunger via the satiety hormone leptin. Blood will be assayed using our standard procedures approximately every six hours.
Ghrelin | 14 days
  The investigators will measure markers of hunger via the hunger hormone ghrelin. Blood will be assayed using our standard procedures approximately every six hours.
Endocannabinoids | 14 days
  The endocannabinoids 2-AG and AEA, as well as non-endocannabinoid N-acylethanolamines (N-oleoylethanolamine [OEA] and N-palmitoylethanolamine [PEA]), and 2-monoacylglycerols (2-oleoylglycerol [2-OG]) via blood. Blood will be assayed using our standard procedures approximately every six hours.
Posture Test Blood Pressure | 14 days
  Standing up after a period of lying down is a large physiological challenge requiring sympathetic activation to maintain perfusion pressure to the brain and void syncope. Participants will be fitted with a 2 lead EKG, a finger cuff for non-invasive BP recordings on a beat-by-beat basis and a sphygmomanometer cuff on the other arm for manual assessment of BP [for cross calibration and safety check]. The finger cuffs will be placed on the non-dominant hand and held in place by an arm sling so that the BP cuffs will be at heart level. BP will be assessed while participants stand up from a semi-recumbent posture and remain standing for ~5min.
Posture Test Heart Rate | 14 days
  Standing up after a period of lying down is a large physiological challenge requiring sympathetic activation to maintain perfusion pressure to the brain and void syncope. Participants will be fitted with a 2 lead EKG, a finger cuff for non-invasive BP recordings on a beat-by-beat basis and a sphygmomanometer cuff on the other arm for manual assessment of BP [for cross calibration and safety check]. The finger cuffs will be placed on the non-dominant hand and held in place by an arm sling so that the BP cuffs will be at heart level. HR will be assessed while participants stand up from a semi-recumbent posture and remain standing for ~5min.
External Temperature Assessment | 14 days
  Skin temperatures (in degrees Celsius) will be continuously assessed using wireless Thermochron iButtons. These iButtons are small (1.6 cm x 0.6 cm), independent temperature sensors and use data loggers enclosed in a watertight stainless-steel package. The iButtons will be taped to the skin with thin, air-permeable adhesive surgical tape in up to 9 different locations and programmed prior to placement via a USB computer interface. Data will be recorded every minute. "Proximal skin temperature" is the averaged skin temperatures of infraclavicular region (mean of left and right) and sternum; "distal skin temperature" is the average skin temperatures of the wrists and ankles.
Internal Temperature Assessment | 14 days
  Temperature data (in degrees Celsius) will also be collected every minute through either rectal thermistors or telemetry pill.The phase of the body temperature rhythm will be determined by the weighted average of the fitted minima of core body temperature data obtained from a single and dual-harmonic fit.
Total Energy Expenditure | 14 days
  Total energy expenditure (TEE) will also be collected across the chronic sleep and circadian disruption protocol by using doubly-labeled water (DLW). DLW is a method based on administration of an oral loading dose of water labeled with both deuterium and oxygen isotope. The tracers quickly equilibrate in the total body water. Deuterium is eliminated from the body in urine only, but the oxygen isotope is eliminated in both urine and carbon dioxide; the difference of the elimination curves is equal to the amount of carbon dioxide expired over the testing period. Urine samples are collected at baseline before the loading dose and again 4-6h after consuming the water on day 1; final urine samples 14 days later.
Changes in Alertness | 14 days
  The investigators will quantify a measure of alertness and hunger to determine the dynamics of acute circadian misalignment and re-entrainment on multiple aspects of waking performance. Alertness will be measured for subjective assessments via a Visual Analog Scale (VAS). The VAS Alert will be performed during sleep inertia testing, which will be the impairment observed immediately upon waking. Sleep inertia testing will occur at ~1, 10, 20, 30, 40, 50, 60, 70, 80, and 90 minutes after waking.
Measuring Mood with POMS | 14 days
  Investigators will measure mood to determine the dynamics of acute circadian misalignment and re-entrainment of waking performance. Mood will be measured by utilizing the POMS questionnaire. The POMS questionnaire is a standard validated psychological test that assesses vigor, fatigue, confusion, anger-hostility, depression, and tension-anxiety by presenting 30 words to participants and requires them to rate how they identify with each word using a numerical value. Each number is associated with a scoring system via a Likert scale (e.g. "Not at All", "A Little", "Moderately", "Quite a Lot" or "Extremely"). These scores are analyzed by a Total Mood Disturbance (TMD) score via the numerical values provided by the participant. Lower scores indicate that a participant has a more consistent or stable mood profile.
  POMS will be administered beginning two hours after waking and repeated every two hours across wakefulness.
Measuring Mood with PANAS | 14 days
  Mood will be additionally investigated by administering the PANAS questionnaire, which is a self-reported measure and consists of different words that describe emotions. There are two scales to this questionnaire, one which measures a positive affect (the ability for a participant to experience positive emotions or interact positively with others), and a negative affect (experiencing negative emotions or interacting negatively with others). Participants will be presented with a questionnaire with 20 words related to emotions and a 5-point Likert scale. Positive affect scores can range from 10-50, with higher scores representing a higher level of positive affect. Negative affect scores can also range from 10-50, and lower scores represent lower levels of negative affect.
  PANAS will be administered beginning two hours after waking and repeated every two hours across wakefulness.
Changes in Degrees of Sleepiness | 14 days
  Investigators will use the Stanford Sleepiness Scale (SSS) for a subjective assessment of sleepiness. The SSS uses a 7-point Likert scale in order to quantify sleepiness at the time of test administration. Values are assigned as follows:
  1. "Feeling active and vital, alert, or wide awake."
  2. "Functioning at a high level, but not at peak; able to concentrate."
  3. "Awake, but relaxed; responsive but not fully alert."
  4. "Somewhat foggy, let down."
  5. "Foggy; losing interest in remaining awake; slowed down."
  6. "Sleepy, woozy, fighting sleep; prefer to lie down."
  7. "No longer fighting sleep, sleep onset soon; having dream-like thoughts."
Changes in Sustained Attention and Reaction Time | 14 days
  Investigators will administer the Psychomotor Vigilance Task (PVT) is a 10 minute, computer-based test in which the participant presses a button as soon as a light appears on the computer screen. This light will appear randomly every few seconds. The main measurements of this task include the mean and median reaction time in milliseconds and sustained attention, as well as false responses. False responses refers to a participant pressing the button before a light is displayed on the computer screen. Individuals who are sleep deprived or are sleep deficit tend to display decreased alertness, declined psychomotor skills, and increased false responses, and therefore have a slower overall reaction time.
  This test will be administered starting two hours after waking and repeated every two hours across wakefulness.
Changes in Cognitive Performance | 14 days
  Cognitive performance will be measured by investigators administering the Digit Symbol Substitution Test (DSST). This is a computer test that presents participants with abstract symbols associated with numbers on a computer screen. The participant must match the symbol that appears on the screen with the corresponding abstract symbol and number. The DSST is a 90 second test and results measured include the total correct and participant errors. Higher scores with fewer errors indicate increased cognitive performance. The DSST will be performed during sleep inertia testing, which will be the impairment observed immediately upon waking. Sleep inertia testing will occur at ~1, 10, 20, 30, 40, 50, 60, 70, 80, and 90 minutes after waking.
Changes in Working Memory | 14 days
  The addition (ADD) task is a 2-digit addition task that will be administered via computer test every 2h to assess working memory. Participants are required to answer as many addition questions as they can within a certain time frame. Results measured include the total correct and participant errors. Higher scores with fewer errors indicate an increased ability to hold information temporarily. The ADD task will be administered two hours after waking and repeated every two hours across wakefulness.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McHill, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No